CLINICAL TRIAL: NCT04633980
Title: Hydrogen Inhalation Therapy in Patients With Moderate Covid-19: Phase-1 Clinical Trial
Brief Title: Hydrogen Therapy in Patients With Moderate Covid-19
Acronym: H2Covid
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 38RC20.277
Record Dates: First submitted 2020-11-16; First posted 2020-11-18 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Covid-19
Keywords: SARS-CoV-2; H2 therapy; ARDS; Inflammation; Oxidative stress
MeSH Terms: conditions — COVID-19; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental)
  Interventions: Drug: Mixture 3,6% H2 in N2 (96.4%)

INTERVENTIONS:
Drug: Mixture 3,6% H2 in N2 (96.4%) — Route of administration: intra-nasal Debit 1L/min, 24h/24h (3 hours withdrawal tolerated) duration of treatment: 24 hours, 3 days and 6 days

SUMMARY:
SARS-CoV-2 is the agent responsible for a new infectious respiratory disease called Covid-19 (for CoronaVirus Disease 2019) which is mainly characterized by potentially severe and fatal lung damage. The severity of the clinical signs associated with this pathology requires the admission to hospital of approximately 20% of patients, 5%-10% of whom will be admitted to intensive care. The most severe cases of this pathology begin with dyspnea which worsens rapidly around the 7th-10th day of the disease into an acute respiratory distress syndrome (ARDS) which requires the patient to be put under mechanical ventilation in the intensive care unit and is responsible for the majority of deaths. Certain biological parameters suggest a massive and brutal release of cytokines (interleukins IL-6, IL-8 and IL-10 mainly) secondary to a syndrome of macrophagic activation mainly in the pulmonary level. Several therapeutic trials aimed at reducing or controlling this immune storm are in progress (anti IL-6 antibodies, anti r IL6 Ab, corticosteroids). Molecular hydrogen acts on the final path of this complex inflammatory cascade by inhibiting the cellular action of reactive oxygen species. Its early use combined with nasal oxygen therapy could prevent this worsening of the respiratory system, so could be likely to limit the risk of overflow of intensive care services during the pandemic and save lives. The aim of this study is to evaluate the safety and the Dose Limiting Toxicity (DLT) of hydrogen therapy delivered by a nasal cannula in addition to conventional oxygen therapy in patients with moderate Covid-19

ELIGIBILITY:
Inclusion Criteria:

1. Patient ≥18 years old
2. Suspicion of SARS CoV-2 infection based on clinical signs AND (positive PCR OR positive serology OR suggestive abnormalities on lung-imaging modalities)
3. Hospitalized patients with SpO2 ≤94% on room air requiring normobaric oxygen therapy with a nasal flow of O2 ≤ 6L / min to reach at least SaO2 ≥ 95%
4. Patient understanding and agreeing to comply with the planned study procedures
5. Patient affiliated with social security or beneficiary of such protection
6. Patient (or his legal representative) who has given his informed consent in writing before the start of any study procedure.

Exclusion Criteria:

1. Pregnant or parturient women
2. Ratio of spontaneous blood ALT/AST> 5 times the normal upper limit.
3. Stage 4 of severe chronic kidney disease or requiring dialysis (i.e. eGFR <30)
4. Early transfer to another hospital within 72 hours.
5. Contraindication to any study drug, including a known allergy
6. Uncontrolled and clinically significant heart disease, such as arrhythmias, angina pectoris or uncompensated congestive heart failure
7. Patients treated in ambulatory care (i.e. not hospitalized)
8. Females of childbearing potential, defined as a premenopausal female capable of becoming pregnant, and not using an highly effective form of birth control.
9. Participant involved in another interventional clinical study
10. Person deprived of liberty by judicial order
11. Person under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-05-23 (Actual)

PRIMARY OUTCOMES:
adverse events | Up to 3 days after the end of H2 therapy
  * observed grade >=4 toxicity from the "Respiratory, thoracic and mediastinal disorders" section of CTCAE v5.0
  * OR observed grade >=3 toxicity from other sections of CTCAE v5.0
  * OR any relevant deterioration in the health of the subject
  * AND at least possibly related with H2

SECONDARY OUTCOMES:
biomarkers of inflammation and oxidative stress. | before and 3 days after the end of H2 therapy
  Serum levels of IL6, IL10, nitrated albumin, and alarmines

CONTACTS AND LOCATIONS:
Overall Officials: Jean Paul Brion, MD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- CHU de Grenoble Alpes, Grenoble, France

REFERENCES:
- [Derived] Salomez-Ihl C, Giai J, Barbado M, Paris A, Touati S, Alcaraz JP, Tanguy S, Leroy C, Lehmann A, Degano B, Gavard M, Bedouch P, Pavese P, Moreau-Gaudry A, Roustit M, Boucher F, Cinquin P, Brion JP. H2 inhalation therapy in patients with moderate COVID-19 (H2COVID): a prospective ascending-dose phase I clinical trial. Antimicrob Agents Chemother. 2024 Aug 7;68(8):e0057324. doi: 10.1128/aac.00573-24. Epub 2024 Jul 17. PMID 39016593